CLINICAL TRIAL: NCT00271037
Title: Pelvic Symptoms and Patient Satisfaction After Colpocleisis for Advanced Pelvic Organ Prolapse
Brief Title: Colpocleisis for Advanced Pelvic Organ Prolapse
Status: Completed | Type: Observational
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Susan Meikle, MD, NICHD
Other Study IDs: 7P01; U01HD041249 (NIH); U10HD041268 (NIH); U10HD041248 (NIH); U10HD041250 (NIH); U10HD041261 (NIH); U10HD041263 (NIH); U10HD041267 (NIH)
Record Dates: First submitted 2005-12-27; First posted 2005-12-29 (Estimated); Last update posted 2011-01-11 (Estimated); Status verified 2010-10

CONDITIONS: Pelvic Organ Prolapse; Stress Urinary Incontinence
Keywords: Pelvic organ prolapse; Stress urinary incontinence; Surgery; Colpocleisis; Urinary retention
MeSH Terms: conditions — Pelvic Organ Prolapse; Urinary Incontinence, Stress; Urinary Retention

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Colpocleisis prolapse repair surgery
Procedure: sling or other to treat or prevent stress incontinence

SUMMARY:
Pelvic organ prolapse occurs when the pelvic organs (e.g., the uterus or bladder) fall or slide down into the vagina. Pelvic organ prolapse can be corrected with surgery. Some types of surgery try to restore the normal anatomy and function of the vagina (i.e., reconstructive surgery). Other surgery repairs the prolapse by essentially closing the vagina (e.g., colpocleisis or colpectomy), thereby leaving a woman unable to have vaginal intercourse in the future. The use of colpocleisis has not been well-studied. The current literature is lacking sufficient studies of colpocleisis to fully understand its risks and benefits for women considering surgery for prolapse. Traditionally, colpocleisis has been restricted to elderly women thought to be poor medical risks for prolonged reconstructive surgery. This study will describe the postoperative course of women who undergo colpocleisis, with particular attention to the persistence or recurrence of urinary incontinence and patient satisfaction after the colpocleisis prolapse surgery.

DETAILED DESCRIPTION:
Pelvic organ prolapse occurs when the pelvic organs (e.g., the uterus or bladder) fall or slide down into the vagina. Pelvic organ prolapse can be corrected with surgery. Some types of surgery try to restore the normal anatomy and function of the vagina (i.e., reconstructive surgery). Other surgery repairs the prolapse by essentially closing the vagina (e.g., colpocleisis or colpectomy), thereby leaving a woman unable to have vaginal intercourse in the future.

The use of colpocleisis prolapse surgery has not been well-studied. The current literature is lacking sufficient studies of colpocleisis to fully understand its risks and benefits for women considering surgery for prolapse. Traditionally, colpocleisis has been restricted to elderly women thought to be poor medical risks for prolonged reconstructive surgery. This study will describe the postoperative course of women who undergo colpocleisis, with particular attention to the persistence or recurrence of urinary incontinence and patient satisfaction after the colpocleisis prolapse surgery.

Women who agree to participate in the study will complete questionnaires before surgery, and at 3 months and 1 year after surgery. Questionnaires include the Pelvic Floor Distress Inventory (PFDI), which includes questions about pelvic symptoms and the level of bother the symptoms cause; the Pelvic Floor Impact Questionnaire (PFIQ), which includes questions about the impact on life activities; and the SF-36, which measures health-related quality of life.

Comparisons: Symptoms that may be related to prolapse, such as urinary incontinence, will be compared in women before and after surgery to see if the surgery provides improvement in those symptoms. In addition, patient satisfaction and health-related quality of life will be studied by making comparisons before and after prolapse surgery repair.

ELIGIBILITY:
Inclusion Criteria:

* Adult women
* Planned colpocleisis or colpectomy surgery for Stage III or Stage IV pelvic organ prolapse
* Able to provide informed consent and complete questionnaire data collection

Exclusion Criteria:

* Planned relocation to nursing home within 3 months of surgery
* Patient preference to maintain coital function after prolapse surgery

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult women undergoing colpocleisis for advanced pelvic organ prolapse (pelvic organ prolapse quantification (POP-Q) stage III-IV)
Sampling Method: Non-Probability Sample
Enrollment: 152 (Actual)
Dates: Start 2004-07; Primary Completion 2007-04 (Actual); Study Completion 2007-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MaryPat FitzGerald, MD, Study Chair — Loyola University
Locations (6):
- United States (6):
  - University of Alabama, Birmingham, Alabama
  - Loyola University, Maywood, Illinois
  - University of Iowa, Iowa City, Iowa
  - Johns Hopkins University, Baltimore, Maryland
  - University of North Carolina, Chapel Hill, North Carolina
  - University of Pittsburgh, Pittsburgh, Pennsylvania

REFERENCES:
- [Background] FitzGerald MP, Richter HE, Siddique S, Thompson P, Zyczynski H; Ann Weber for the Pelvic Floor Disorders Network. Colpocleisis: a review. Int Urogynecol J Pelvic Floor Dysfunct. 2006 May;17(3):261-71. doi: 10.1007/s00192-005-1339-9. Epub 2005 Jun 28. PMID 15983731
- [Result] Fitzgerald MP, Richter HE, Bradley CS, Ye W, Visco AC, Cundiff GW, Zyczynski HM, Fine P, Weber AM; Pelvic Floor Disorders Network. Pelvic support, pelvic symptoms, and patient satisfaction after colpocleisis. Int Urogynecol J Pelvic Floor Dysfunct. 2008 Dec;19(12):1603-9. doi: 10.1007/s00192-008-0696-6. Epub 2008 Aug 9. PMID 18690402
- [Result] Gutman RE, Bradley CS, Ye W, Markland AD, Whitehead WE, Fitzgerald MP; Pelvic Floor Disorders Network. Effects of colpocleisis on bowel symptoms among women with severe pelvic organ prolapse. Int Urogynecol J. 2010 Apr;21(4):461-6. doi: 10.1007/s00192-009-1062-z. Epub 2009 Dec 4. PMID 19960182
- [Derived] Barber MD, Chen Z, Lukacz E, Markland A, Wai C, Brubaker L, Nygaard I, Weidner A, Janz NK, Spino C. Further validation of the short form versions of the Pelvic Floor Distress Inventory (PFDI) and Pelvic Floor Impact Questionnaire (PFIQ). Neurourol Urodyn. 2011 Apr;30(4):541-6. doi: 10.1002/nau.20934. Epub 2011 Feb 22. PMID 21344495
- See also: Website of the National Institute of Child Health and Human Development, which funds the Pelvic Floor Disorders Network — http://www.nichd.nih.gov